CLINICAL TRIAL: NCT02369302
Title: An Open-label, Randomized, 6-Sequence, 3-Period Crossover Study to Evaluate a Drug Interaction Between DWC20141 and DWC20142 in Healthy Adult Subjects
Brief Title: Pharmacokinetics and Drug Interaction Study Between DWC20141 and DWC20142 in Healthy Male Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Daewoong Pharmaceutical Co. LTD. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: DW_DWJ1367001
Record Dates: First submitted 2015-02-17; First posted 2015-02-23 (Estimated); Last update posted 2016-03-01 (Estimated); Status verified 2016-02

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- DWC20141 (Experimental): multiple dose of DWC20141
  Interventions: Drug: DWC20141
- DWC20142 (Experimental): multiple dose of DWC20142
  Interventions: Drug: DWC20142
- DWC20141+DWC20142 (Experimental): multiple dose of DWC20141 and DWC20142
  Interventions: Drug: DWC20141, DWC20142

INTERVENTIONS:
Drug: DWC20141 — Tablet
  Arms: DWC20141
Drug: DWC20142 — Tablet
  Arms: DWC20142
Drug: DWC20141, DWC20142 — Tablet
  Arms: DWC20141+DWC20142

SUMMARY:
The purpose of this study is to evaluate the pharmacokinetics profile and drug-drug interaction between DWC20141 and DWC20142 in healthy adult subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy adult male volunteers aged 19 to 45 years
2. A sybject who has judged to be healthy by the investigator to participate in this study based on screening result
3. A subject who provided written informed consent to participate in this study and cooperative with regared to compliance with study related constraints

Exclusion Criteria:

1. A subject with sign or symptoms or previously diagnosed disease of liver, digestive system, cardiovascular, kidney, respiratory, endocrinology, neurology, immune system, hematology, and psychology function or other significant disease and history.
2. A subject who shows the following result in clinical laboratory test

   * AST, ALT > 1.25 times of the upper limit of normal range
   * PR ≥ 210 msec
   * QRS ≥ 120 msec
   * QT ≥ 500 msec
   * QTcF ≥ 500 msec
3. Subject who has taken other clinical medication from another clinical trial within 3-months period prior to the first administration of the study medication.

Ages: 19 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2015-01; Primary Completion 2015-03 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Cmax,ss | Multiple blood sample will be collected for 24 hours after last dosing in each of the periods
AUCtau | Multiple blood sample will be collected for 24 hours after last dosing in each of the periods

SECONDARY OUTCOMES:
Cmin,ss | Multiple blood sample will be collected for 24 hours after last dosing in each of the periods
Tmax | Multiple blood sample will be collected for 24 hours after last dosing in each of the periods
t1/2 | Multiple blood sample will be collected for 24 hours after last dosing in each of the periods
Metabolic Ratio | Multiple blood sample will be collected for 24 hours after last dosing in each of the periods

CONTACTS AND LOCATIONS:
Overall Officials: Eun-Young Kim, Professor, Principal Investigator — BUSAN PAIK HOSPITAL
Locations (1):
- Inje University College of Medicine Busan Paik Hospital, Busan, Busanjin-gu, South Korea